CLINICAL TRIAL: NCT06477536
Title: A Phase IIb, Long-Term Extension Study to Evaluate the Safety and Efficacy of HB0034 in the Treatment of Adult Subjects With Generalized Pustular Psoriasis
Brief Title: Long-Term Safety and Efficacy of HB0034 in Subjects With Generalized Pustular Psoriasis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB0034-05
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-09

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HB0034 (Experimental): single-arm and all the patients would receive HB0034 300mg i.v. every other four weeks
  Interventions: Drug: HB0034

INTERVENTIONS:
Drug: HB0034 — 300mg, i.v. Q4W
  Other Names: Anti-IL-36R antibody,Recombinant Humanized anti-IL-36R Monoclonal antibody

SUMMARY:
This is a Phase IIb, long term extension study to evaluate the safety and efficacy of HB0034 in adult subjects with generalized pustular psoriasis (GPP).

DETAILED DESCRIPTION:
This study will also evaluate the pharmacokinetic (PK) profile of HB0034 and explore the immunogenicity of HB0034 in subjects with GPP

ELIGIBILITY:
Inclusion Criteria:

* Patients participated in the preceding placebo-controlled Phase 2 study （HB0034-04）and completed at least the Week 12 visit of the HB0034-04 study
* Subject must be a candidate for prolonged GPP treatment according to the Investigator's judgment
* Men and women of reproductive age who have no parenting plans and are willing to use reliable contraception during the study period and for 6 months after the last dose of the study drug;
* Patients who fully understand and voluntarily sign an ICF, and are willing and able to follow clinical study and subsequent visit schedules

Exclusion Criteria:

* Patients who are experiencing GPP flare

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints include the proportion of subjects with TEAEs | 0-24 weeks
  The safety assessment includes monitoring for AEs, SAEs (including SAEs related to protocol procedures from signing of ICF until before the first dose of the study drug) from the first dose of the study drug to end of study (EOS) , as well as changes from baseline in laboratory tests, vital signs, physical examination, and 12-lead electrocardiogram (ECG).

SECONDARY OUTCOMES:
The recurrence of GPP flare during the study | 0-24 weeks
  The Proportion of patients who have at least once GPP flare during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, PhD, Principal Investigator — Peking University People's Hospital (PKUPH)
Locations (3):
- China (3):
  - Peking University People's Hospital (PKUPH), Beijing
  - Peking University People's Hospital, Beijing
  - The Second affiliated Hospital zhejiang University School of Medicine, Hangzhou